CLINICAL TRIAL: NCT06472258
Title: Efficacy of Only IV Artesunate Versus IV Artesunate Plus IV Quinine in the Treatment of Severe Malaria in Children: A Comparative Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RESnTEC, Institute of Research (Other)
Responsible Party: Principal Investigator, Muhammad Aamir Latif, Investigator, RESnTEC, Institute of Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DGKhan
Record Dates: First submitted 2024-06-14; First posted 2024-06-25 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — Artesunate; Quinine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IV Artesunate Group (Experimental): IV Artesunate with weight appropriate dosage on 0, 12, 24 and 48 hours, and continued 12 hourly for a maximum duration of seven days. Each dose diluted in normal saline given as infusion.
  Interventions: Drug: IV Artesunate
- Combination Group (Experimental): IV Artesunate with weight appropriate dose on 0, 12, 24 and 48 hours, plus IV Quinine hydrochloride in accordance to weight with loading dose 20mg salt/kg in 10% dextrose infusion followed by 10mg salt/kg infusion 8 hourly for 2 days and for 12 hourly onwards for a maximum of 7 days.
  Interventions: Drug: IV Artesunate; Drug: IV Quinine Hydrochloride

INTERVENTIONS:
Drug: IV Artesunate — IV artesunate with a weight-appropriate dosage at 0, 12, 24, and 48 hours and continued 12-hourly for a maximum duration of seven days, with each dose diluted in normal saline and given as an infusion.
  Other Names: Artesunate
Drug: IV Quinine Hydrochloride — IV Quinine hydrochloride in accordance to weight with loading dose 20mg salt/kg in 10% dextrose infusion followed by 10mg salt/kg infusion 8 hourly for 2 days and for 12 hourly onwards for a maximum of 7 days.
  Other Names: Artesunate plus IV Quinine Hydrochloride
  Arms: Combination Group

SUMMARY:
The WHO recommends artesunate as the drug of choice for the treatment of severe malaria. However, the efficacy of this single drug as compared to the combined drug regimen remained questionable, and the clinical response was considered delayed or inappropriate. Therefore, this research intended to evaluate the efficacy of only IV artesunate versus IV artesunate plus IV quinine in the treatment of severe malaria in children. The findings of the study would be helpful knowing whether the two drugs, when given together, have considerable benefit over single-drug therapy when given for the same.

ELIGIBILITY:
Inclusion Criteria:

Children admitted to the emergency department with the diagnosis of severe malaria.

Exclusion Criteria:

Children with chronic kidney disease, chronic liver disease, immunosuppressive disorders, hematological disorders, malignancies, and congenital heart disease.

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 104 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Efficacy measurement between IV Artesunate and IV Artesunate plus IV Quinine Hydrochloride | Seven days
  The outcome was measured in the number of hours elapsed for an individual to become fever-free.

CONTACTS AND LOCATIONS:
Locations (1):
- Allama Iqbal Teaching Hospital, Dera Ghazi Khan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
It can be shared on a reasonable request made to primary investigators.